CLINICAL STUDY OF BIOLOGICAL AND MECHANICAL COMPLICATIONS IN SINGLE IMPLANT PROSTHESIS WITH OR WITHOUT INTERMEDIATE ABUTMENT

March 24th 2022

## INFORMED CONSENT FORM TO PARTICIPATE IN THE STUDY

| Mr/Mrs: |
|---|
| Date of birth: |
| ID: |
| Home: |
| DECLARES |
| I will participate in the study that bears the name: |
| I will do it voluntarily. |
| It has been explained to me that: |
| 1 The main purpose of the study is to analyze the possible complications that may appear in the rehabilitation treatment with implants that I am going to receive. |
| 2 All my data will be protected in compliance with the Law of Protection of Personal Data, Organic Law 15/1999, of 13December, Personal Data Protection. |
| I have understood the explanations that have been provided to me in clear language |
| and simple, and the doctor who has treated me has allowed me to carry out all the |
| observations and has clarified all the doubts that I have raised. |
| Likewise, I confirm that the explanations and my questions have been made with prior |
| to carrying out the treatment, and that I have sufficient time to reconsider the information |
| received and be able to make further observations if so deemed it necessary. |
| I also understand that at any time and without giving any explanation, I can revoke the |
| consent that I now give. |
| Therefore, I state that I am satisfied with the information received and that |
| I understand the scope and risks of the study, and under such conditions. |
| I <b>CONSENT</b> to be included in the study in which I am going to take part. |
| In León, at of 20 |
| Signed: The volunteer. |

I have understood the explanations that have been provided to me in clear language and simple, and the doctor who has treated me has allowed me to carry out all the observations and has clarified all the doubts that I have raised.

I also understand that at any time and without giving any explanation, I can revoke the consent that I now give.

| Therefore, I state that I am satisfied with the information received that |
|---------------------------------------------------------------------------|
| I understand the scope and risks of the study, and under such conditions. |
| I CONSENT that they can pour results regarding the questionnaire that |
| I will reply below. |
| In , at from of 20 |
| Signed: The volunteer. |